CLINICAL TRIAL: NCT00001239
Title: Combination Chemotherapy (FLAC) Combined With Granulocyte-Macrophage Colony Stimulating Factor in Locally Advanced and Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 890119; 89-C-0119
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-04

CONDITIONS: Breast Cancer; Breast Neoplasms
Keywords: 5-Fluorouracil; Adriamycin; Breast Carcinoma; Leucovorin; Phase II
MeSH Terms: conditions — Breast Neoplasms | interventions — Granulocyte-Macrophage Colony-Stimulating Factor

INTERVENTIONS:
Drug: FLAC with GM-CSF

SUMMARY:
To evaluate a dose intensive chemotherapy regimen for the treatment of locally advanced and metastatic breast cancer using granulocyte-macrophage colony-stimulating factor (GM-CSF) to ameliorate chemotherapy-induced toxicity. Combination chemotherapy consists of Flurouricil, Leucovorin, Adriamycin, and Cytoxan (FLAC) which will be given every 21 days for 10 cycles. This protocol will replace the phase I study of this regimen (MB-232/88-C-0207) which found the MTD of this regimen to be at the first dose level. This is a phase II study to determine response rates of this regimen in advanced breast cancer.

DETAILED DESCRIPTION:
To evaluate a dose intensive chemotherapy regimen for the treatment of locally advanced and metastatic breast cancer using granulocyte-macrophage colony-stimulating factor (GM-CSF) to ameliorate chemotherapy-induced toxicity. Combination chemotherapy consists of Flurouricil, Leucovorin, Adriamycin, and Cytoxan (FLAC) which will be given every 21 days for 10 cycles. This protocol will replace the phase I study of this regimen (MB-232/88-C-0207) which found the MTD of this regimen to be at the first dose level. This is a phase II study to determine response rates of this regimen in advanced breast cancer.

ELIGIBILITY:
All stage III or clinical T3N0 or TxN2 patients must have a histologically documented diagnosis of breast carcinoma and evaluate disease in the breast or axilla.

Patients with stage III must enter this protocol within 12 weeks of the initial diagnosis.

Patients with Stage IV (metastatic) breast cancer must have histologically proven diagnosis and must have evaluate disease. Patients with bone-only disease may be considered eligible after discussion with Dr. Kenneth Cowan.

For Stage III disease, there must be no history of prior cytotoxic therapy.

Stage IV patients will be eligible if they have had prior adjuvant chemotherapy and/or hormonal therapy provided the regimen did not included adriamycin. Patients will also be eligible if they have been treated with one prior Phase I or II single chemotherapy agent on a Medicine branch protocol. Patients who have had prior radiation therapy may be eligible providing there was not extensive radiation to the cardiac area.

There must be no history of previous malignancy except for cured non-melanoma skin cancer (basal cell carcinoma) and cervical cancer in situ.

Performance status (Karnofsky scale) must be greater than 70.

WBC count greater than 4000/mm3 and platelet count 100,000/mm3, unless there is evidence of bone marrow involvement with tumor.

Liver function tests (SGOT, Alk. Phosph., and T. Bilil) should be less than 1.5 times the upper limits of normal, and serum creatinine should be less than 1.7 or creatinine clearance should be greater than 45 ml/min unless these abnormalities are due to tumor involvement.

The patient must give informed consent.

No pregnant patients may be entered on this study; all patients should be informed about the need for contraception.

No history of other malignant neoplasms except for curatively treated basal cell skin cancer or surgically cured carcinoma of the cervix in situ.

Patients must not be in poor medical or psychiatric risks because of nonmalignant systemic disease which would preclude them being subjected to any treatments in this protocol.

Patients with a history of cardiac disease must have a normal ejection fraction by MUGA Scan and have no angina.

Must not have evidence of CNS metastasis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 1989-07; Study Completion 2001-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Swain SM, Sorace RA, Bagley CS, Danforth DN Jr, Bader J, Wesley MN, Steinberg SM, Lippman ME. Neoadjuvant chemotherapy in the combined modality approach of locally advanced nonmetastatic breast cancer. Cancer Res. 1987 Jul 15;47(14):3889-94. PMID 3036348
- [Background] Antman K, Gale RP. Advanced breast cancer: high-dose chemotherapy and bone marrow autotransplants. Ann Intern Med. 1988 Apr;108(4):570-4. doi: 10.7326/0003-4819-108-4-570. PMID 3279894
- [Background] Clark SC, Kamen R. The human hematopoietic colony-stimulating factors. Science. 1987 Jun 5;236(4806):1229-37. doi: 10.1126/science.3296190.